CLINICAL TRIAL: NCT04395586
Title: Clinical Presentations, Microbiology, Antibiotic Resistance Patterns and Management Outcomes of Culture-proven Infection Among Adolescent and Adult in A Tertiary Hospital in Saudi Arabia
Status: Withdrawn | Type: Observational
Why Stopped: Due to COVID-19 panemic
Sponsor: Aseer Central Hospital (Other Government)
Responsible Party: Principal Investigator, Abdullah M. Algarni, Family medicine senior registrar, Aseer Central Hospital
Other Study IDs: ACH-1
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Culture-proven Infection
MeSH Terms: interventions — Culture Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Study will include a sample from blood, cerebrospinal fluid, intra-articular fluid, peritoneal fluid, pleural fluid, sputum, tissue (e.g., skin, bone, and cartilages), and urine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Culture-proven infected patients
  Interventions: Other: Culture

INTERVENTIONS:
Other: Culture — Culture

SUMMARY:
The characteristics of patients as well as microbiologic profile of culture-proven infection will be studies in conjunction with clinical outcome within 28-days

ELIGIBILITY:
Inclusion Criteria:

* Any individual aged ≥13 year old requested for him/her bacterial/fungal culture.
* Able to provide a written informed consent.

Exclusion Criteria:

* Age <13 years old.
* Unable/unwilling to provide a written informed consent.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any individual aged ≥13 year old requested for him/her bacterial/fungal culture.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28 days
  All-cause and disease specific mortality

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah M Algarni, MBBS, Principal Investigator — Aseer Central Hospital

IPD SHARING:
Plan to Share IPD: No